CLINICAL TRIAL: NCT00004987
Title: Intraperitoneal Dextrin Sulfate in Patients With Advanced HIV Disease: A Phase I Trial
Brief Title: Treatment of Advanced AIDS Patients With Dextrin Sulfate
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Steinhart Medical Associates (Other)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 309A
Record Dates: First submitted 2000-03-16; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-06

CONDITIONS: HIV Infections
Keywords: Anti-HIV Agents; Viral Load; dextrin 2-sulfate; Infusions, Parenteral
MeSH Terms: conditions — HIV Infections | interventions — dextrin 2-sulfate

INTERVENTIONS:
Drug: Dextrin 2-sulfate

SUMMARY:
The purpose of this study is to look at the safety and effectiveness of dextrin sulfate in AIDS patients who have failed conventional anti-HIV treatment.

DETAILED DESCRIPTION:
Patients have intraperitoneal (IP) catheter placement done at study entry. Infusion with the carrier vehicle (icodextrin 4%) begins 2 weeks later, and 2 days after that, treatment with dextrin sulphate (DS) commences. DS is given three times per week. A nurse delivers initial treatments and the patient and caregiver will be trained to give subsequent treatments until DS has been given a total of 8 weeks. Patient evaluations are done regularly during treatment and observation continues for 24 weeks.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this trial if they:

* Are HIV-positive.
* Have been diagnosed with AIDS and are under treatment to prevent opportunistic (AIDS-related) infection.
* Have had a CD4 cell count greater than 50 microL for at least the past 3 months.
* Have had a viral load of at least 50,000 copies/ml for at least the past 3 months.
* Have used up all other treatment options.
* Are able to understand and give written consent.

Exclusion Criteria

Patients may not be eligible for this trial if they:

* Have been in any other study in the 6 weeks before beginning this study.
* Have an active, opportunistic infection or other infection.
* Have any other long-term medical condition or nervous disorder that might make it difficult for them to finish the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-10

CONTACTS AND LOCATIONS:
Locations (1):
- Steinhart Medical Associates, Miami, Florida, United States